CLINICAL TRIAL: NCT03944837
Title: Congenital Heart Disease (CHD): Hemodynamic Effects of Acute Maternal Hyperoxygenation in the Fetus
Brief Title: Acute Maternal Hyperoxygenation in CHD
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: The Hospital for Sick Children (Other)
Responsible Party: Principal Investigator, Edgar Jaeggi, Primary Investigator, The Hospital for Sick Children
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1000062939
Record Dates: First submitted 2019-04-29; First posted 2019-05-10 (Actual); Last update posted 2024-01-31 (Actual); Status verified 2024-01

CONDITIONS: Congenital Heart Disease
Keywords: Acute maternal hyperoxygenation; Echocardiography; MRI
MeSH Terms: conditions — Heart Defects, Congenital | interventions — nitrox

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Severe fetal congenital heart disease (CHD) (Experimental): Mothers whose fetuses have a diagnosis of CHD will be exposed to 10-15 L/minute of oxygen while undergoing echocardiogaphy and MRI scanning
  Interventions: Other: Oxygen gas

INTERVENTIONS:
Other: Oxygen gas — Transient maternal oxygen administration during echocardiographic and MRI imaging

SUMMARY:
Congenital heart disease (CHD) is predominantly detected before birth. Using echocardiography and MRI, this study will determine whether acute exposure to maternal hyperoxygenation (MH) leads to measurable increases in fetal cerebral oxygenation from baseline in fetuses with CHD. The study aims to determine whether MH could be used as a chronic in-utero treatment strategy to promote brain growth/maturation to birth and to improve postnatal neurodevelopmental outcomes, and identify the types of CHD most likely to benefit from chronic MH.

DETAILED DESCRIPTION:
This study determines the impact of administering oxygen to mother during the later part of pregnancy on cerebral oxygen delivery in fetuses who were identified with severe forms of Congenital Heart disease (CHD) including the following groups:

* Group 1: Single ventricular (SV) lesions, including hypoplastic left heart syndrome (HLHS); pulmonary atresia with intact ventricular septum (PA/IVS); tricuspid atresia (TA); unbalanced AV septal defect (AVSD); double inlet ventricle (DILV); and severe form of Ebstein's anomaly (EA with pulmonary atresia) of the tricuspid valve; and
* Group 2: Tetralogy of Fallot (TOF),including TOF-like double outlet right ventricle (DORV), pulmonary atresia with ventricular septal defect (PA/VSD)
* Group 3: Bi-ventricular lesions with transposition of the great arteries (TGA), including DORV with TGA

Children with severe CHD experience challenges in multiple developmental domains, impacting executive function, memory, language, and other aspects of cognitive and motor function. It is now well established that brain growth and development are adversely affected by CHD and it is increasingly clear that central nervous system changes that occur in the third trimester play a particularly important role in the pathogenesis of adverse neurodevelopmental outcomes.

Supplemental maternal oxygen will used in the last trimester for a short period of time (acute MH) in pregnant mothers carrying babies with CHD to briefly increase fetal oxygen levels to those reached in the newborn with spontaneous breathing. This study will examine whether and to what degree acute MH will improve the cerebrovascular oxygenation. The rate and duration of MH (10 to 15L/min by mask for up to 30-45 minutes/test) is considered to be safe to the mother and her fetus. Both fetal echocardiography and fetal MRI will be used to determine the effects of acute MH on the fetal-placental circulation and will determine in fetuses with CHD whether acute exposure to MH leads to measurable increases in fetal cerebral oxygenation from baseline. Thus it could potentially become useful as a chronic in-utero treatment strategy to promote brain growth/maturation to birth and to improve postnatal neurodevelopmental outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant mothers ≥18 years of age
* Written maternal informed consent
* Fetal diagnosis of one of the CHDs (1-3) as listed below and intention of active treatment after birth:

  1. Single ventricular (SV) lesions: hypoplastic left heart syndrome (HLHS); pulmonary atresia with intact ventricular septum (PA/IVS); tricuspid atresia (TA); unbalanced AV septal defect (AVSD); double inlet ventricle (DILV); and severe form of Ebstein's anomaly (EA) of the tricuspid valve associated with functional or anatomical right outflow obstruction. HLHS will include aortic stenosis with mitral stenosis, aortic atresia with mitral stenosis or mitral atresia. Pulmonary or aortic obstruction is defined as a condition with minimal or absent antegrade flow across the respective valve. Severe forms of EA is defined as lesion without anterograde pulmonary flow in the setting of severe tricuspid regurgitation.
  2. Bi-ventricular lesions with right ventricular outflow tract obstruction (BV/RVOTO); tetralogy of Fallot (TOF), TOF-like double outlet right ventricle (DORV), and pulmonary atresia with ventricular septal defect (PA/VSD).
  3. Bi-ventricular lesions with transposed great arteries (TGA w/ VSD; TGA w/o VSD; DORV with TGA)

Exclusion Criteria:

* Termination of pregnancy
* Unusual CHDs (e.g. EA with circular shunt, TOF with AVSD, and TOF with absent pulmonary valve syndrome, TGA associated with moderate- severe outflow tract obstruction
* Complex cardiac condition (e.g poor fetal cardiac function and/or fetal hydrops, fetal arrhythmia such as frequent premature atrial beats, abnormal baseline heart rate (<110 bpm; > 160 bpm) in the third trimester)
* Major non-cardiac lesions and major genetic abnormalities affecting brain size and development
* Significant maternal co-morbidities that precludes a fetal MRI (e.g. significant obesity, claustrophobia)
* Multiple pregnancy

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2019-04-26 (Actual); Primary Completion 2024-08-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Characterize the hemodynamic effects of acute MH on fetuses with a) SV lesions and biventricular anomalies b) with TOF and c) with TGA. | Outcome measure obtained during hyperoxygenation while undergoing echocardiography and MRI
  The affect MH has on the cerebral oxygenation from baseline for each type of CHD will be characterized using the MRI variables of cerebral oxygen delivery (cDO2) and cerebral oxygen consumption(cVO2) , which are calculated using fluximetry measurements (ml/min/m2) and the oxymetry of the ascending aorta and the superior vena cava

SECONDARY OUTCOMES:
Determine the pulmonary and placental vascular response to acute MH for each CHD | Outcome measure obtained during hyperoxygenation while undergoing echocardiography and MRI
  The pulmonary and placental vascular response to acute MH for each CHD type will be measured using the placenta T2 star variable and the variables related to main pulmonary artery and branch pulmonary artery flow. Pulmonary vaso-reactivity to oxygen by echocardiography defined by a decrease the branch PA PI of ≥10%.

OTHER OUTCOMES:
Assess the relationship between fetal brain volumes and cerebral oxygen delivery | Outcome measure obtained during hyperoxygenation while undergoing echocardiography and MRI
  The fetal brain volumetry (mL) and rate of cerebral oxygen delivery (cDO2 ml/min/m2) at the time of the baseline fetal MRI will be compared
To compare the prenatal measurement of placenta and the growth in body and brain size at birth. | Date of echocardiography/MRI to the date of the infant's birth, when the birth weight, height and head circumference data become available.
  The placental measurement by MRI will be correlated with head circumference and body weight at birth.

CONTACTS AND LOCATIONS:
Overall Officials: Edgar Jaeggi, MD, FRCP(C), Principal Investigator — The Hospital for Sick Children; Mike Seed, MBBS, Principal Investigator — The Hospital for Sick Children
Locations (1):
- The Hospital for Sick Children, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No